CLINICAL TRIAL: NCT04984369
Title: An Open, Multicenter Phase II Clinical Study to Evaluate Safety and Efficacy of HLX208 (BRAF V600E Inhibitor) Combined With Cetuximab in Patients With Metastatic Colorectal Cancer (mCRC)
Brief Title: The Efficacy of HLX208 (BRAF V600E Inhibitor) With Cetuximab for Metastatic Colorectal Cancer (mCRC) With BRAF V600E Mutation After First-line Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX208-mCRC201（BECOMES）
Record Dates: First submitted 2021-07-27; First posted 2021-07-30 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: CRC
MeSH Terms: interventions — CCT239065; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Never use other BRAF inhibitor therapy (Experimental): Never use other BRAF inhibitor therapy
  Interventions: Drug: HLX208; Drug: Cetuximab Injection [Erbitux]
- PD after other BRAF inhibitor therapy N=5~40 (Experimental): PD after other BRAF inhibitor therapy
  Interventions: Drug: HLX208; Drug: Cetuximab Injection [Erbitux]
- SD but intolerant after other BRAF inhibitor therapy (Experimental): SD but intolerant after other BRAF inhibitor therapy
  Interventions: Drug: HLX208; Drug: Cetuximab Injection [Erbitux]

INTERVENTIONS:
Drug: HLX208 — HLX208 450mg bid po OR 600mg bid po OR 900mg bid po
  Other Names: BRAF V600E inhibitor
Drug: Cetuximab Injection [Erbitux] — Cetuximab 500 mg/m2 IV Q2W

SUMMARY:
An open, multicenter phase II clinical study to evaluate safety and efficacy of HLX208 (BRAF V600E inhibitor) combined with cetuximab for metastatic colorectal cancer (mCRC) with BRAF V600E Mutation after first-line treatment

ELIGIBILITY:
Inclusion Criteria:

* Age>=18Y
* Good Organ Function
* Expected survival time ≥ 3 months
* Metastatic/recurrent advanced BRAF+ mCRC that have been diagnosed histologically and have failed first line treatment
* ECOG score 0-1;

Exclusion Criteria:

* arm 1 ： Previous treatment with BRAF inhibitors or MEK inhibitors
* Symptomatic brain or meningeal metastases (unless the patient has been on > treatment for 3 months, has no evidence of progress on imaging within 4 weeks prior to initial administration, and tumor-related clinical symptoms are stable).
* Active clinical severe infection;
* A history of other malignancies within two years, except for cured carcinoma in situ of the cervix or basal cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 2 years
  Objective response rate(assessed by independent radiological review committee (IRRC) based on the RECIST Version 1.1)

SECONDARY OUTCOMES:
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 2 years]
  Progression-free survival (PFS) (assessed by IRRC and the investigator as per RECIST v1.1 )
OS | from the date of first dose until the date of death from any cause，assessed up to 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Affiliated Oncology Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No